CLINICAL TRIAL: NCT04821193
Title: Comparison of the Effects of 5% NaHCO3, 2% Chlorhexidine Gluconate and 70% Alcohol for Prevention of Infections Related to Catheter Applications in Children.
Brief Title: Comparison of the Effects of 5%NaHCO3, 2%CHG and 70%Alcohol in the Prevention of Infections Related to Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aysegul Simsek, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Antiseptic
Record Dates: First submitted 2021-03-18; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Disinfectant Dye Adverse Reaction; Catheter-Related Infections; Nursing Caries; Children, Only; Skin Lesion; Chlorhexidine Adverse Reaction; Catheter
Keywords: Antiseptic; Intravenous catheterization; Catheter-related infection; Chlorhexidine gluconate; Sodium bicarbonate
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Intervention Model Description: Single blind Randomized controlled Experimental
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental Group 1 (Experimental): Cleansing the skin with an antiseptic solution before intravenous catheterization Skin antisepsis with 5% NaHCO3 water solution group Grup number: 20
  Interventions: Drug: Skin antisepsis with 5% NaHCO3 water solution
- Experimental Group 2 (Experimental): Cleansing the skin with an antiseptic solution before intravenous catheterization Skin antisepsis with 2% Chlorhexidine Gluconate solution group Grup number: 21
  Interventions: Drug: Skin antisepsis with 2% Chlorhexidine Gluconate solution
- Control Group (No Intervention): Cleansing the skin with an antiseptic solution before intravenous catheterization Skin antisepsis with 70% Alcohol solution group Grup number: 21

INTERVENTIONS:
Drug: Skin antisepsis with 5% NaHCO3 water solution — In-vitro analysis of the solutions was done first. Then solutions were applied, and peripheric intravenous catheter was installed
  Other Names: Disinfectant drugs; Chemical substance
  Arms: Experimental Group 1
Drug: Skin antisepsis with 2% Chlorhexidine Gluconate solution — In-vitro analysis of the solutions was done first. Then solutions were applied, and peripheric intravenous catheter was installed
  Other Names: Disinfectant drugs; Chemical substance
  Arms: Experimental Group 2

SUMMARY:
Intravenous catheters have become one of the indispensable tools of modern medicine. Peripheric intravenous catheters facilitate the work of healthcare professionals in the treatment phase, especially in diagnostic procedures. Intravenous catheters cause microorganisms to enter the bloodstream by damaging the skin, which is the body's first defense barrier. In this case, it causes infections, sepsis, an increase in mortality and morbidity rates, prolongation of hospital stay, increase in antibiotic use, and medical expenses. The density of the skin flora in the area where the catheter will be inserted is a major risk factor for infection.To prevent complications associated with peripheric intravenous catheters; Performing the procedure in line with the principles of surgical asepsis and following the correct follow-up are among the most important measures that the nurse should take. Also, the child and the parents should be prepared for the procedure and the appropriate environment should be provided. Along with correct catheter placement and care, antisepsis of the cannula placement area is among the indicators of nursing care.

As well as the effectiveness and safety of skin disinfectants, topical absorption, lack of toxic effect, local and irritation effect are also important. Solutions with 5% NaHCO3 have recently come to the fore as antiseptic agents. When the literature is examined, it has not been found that there are very few studies on this solution and it is used in skin antisepsis before peripheral intravenous catheterization in children. This study was planned as a randomized controlled experimental design to determine the effectiveness of 5% NaHCO3 water solution in catheter site cleaning in pediatric patients by comparing it with the most commonly used antiseptic agents and to monitor the development of catheter-related infections.

DETAILED DESCRIPTION:
Intravenous therapy is one of the basic elements of modern health care. IV routes provided through catheters for pediatric patients are necessary for primary and secondary health and increase the possibility of mortality and morbidity depending on the treatment given and the factors of the patient. As in every invasive application, there are problems regarding the use of catheters, which is a minimal surgical procedure, and perhaps the most important of these is catheter-related infections.

CRI's are defined as the accompanying of both local (redness around the catheter, increased temperature, discharge, drainage, tenderness, edema) and systemic (fever, chills, changes in laboratory tests) infection findings in patients and is an important complication for children. is happening. The increase in prevalence varies among patients, as well as between cities and countries, and is among the top three among hospital-associated infections.

Although there are many studies on infections related to the use of a peripheric intravenous catheters in adult patients, it is reported that this issue is not addressed much in children. It is thought that there is no standardization regarding peripheric intravenous catheters management in the studies conducted.

Since the risk factors for infection such as body weight, concomitant chronic disease, characteristics of the catheter used and the drug administered, presence of interconnection for pediatric patients are different from adults, catheter-related infections in the pediatric age group requires a separate discussion. It cannot be denied that the main step in the prevention of catheter-related infections is the management of peripheric intravenous catheters and determining an appropriate skin antiseptic is a part of this.

In Children, 70% Alcohol, 2% Chlorhexidine Gluconate, 1% Octenidine, and 10% Povidone-iodine type antiseptics are commonly used for skin antisepsis. Sodium bicarbonate (NaHCO3) solutions are used in different areas such as oral hygiene and dental care in the world and our country, and side effects are not reported. There is limited information in the literature regarding its use as a skin antiseptic, and it is seen that this information belongs to the adult age group. There is no data on the child age group.

In this study, which was planned in two stages to determine the effectiveness of the use of sodium bicarbonate as a skin antiseptic in the prevention of catheter-related infections, the effectiveness of the antiseptics used in the first stage was evaluated in the laboratory environment against the most common microorganisms in the skin flora, and in the second stage, the use of these antiseptic solutions in skin cleansing in pediatric patients before the peripheric intravenous catheters procedure their effectiveness has been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 1-18
* Having inpatient treatment in pediatric clinics
* No previous history of catheter-related infections
* No history of systemic infection
* Absence of immunological disease
* Not using antibiotherapy
* No scar/scar tissue on the skin in the catheterization area

Exclusion Criteria:

* Being an inpatient who does not need intravenous treatment
* Finding an infection
* Having a chronic skin disease
* Having a history of allergies
* Being a newborn

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
The effectiveness of the solutions - In-vitro analysis | One months
  Effectiveness in the laboratory: The efficacy of the solutions on the most common bacteria on the skin was tested in the laboratory.
  Analysis of solutions to be used in Laboratory Environment (In vitro): 5% NaHCO3 water solution, 2% KHG solution and 70% Alcohol solution to be used in the catheterization process were studied in the laboratory with the microbiologist in the blood, Müller Hinton agar with disk diffusion method.
  The diameter of the discs used is 9 mm. Microorganisms are clinical isolates. As a result, they are the inhibition zones recorded.

SECONDARY OUTCOMES:
The effectiveness of the solutions - Practice | Five months
  Before the process, the solutions were prepared by the researcher weekly in the laboratory. The solution to be administered to the patients was determined by randomization.
  In the units where the study was conducted, peripheral intravenous catheters were placed in the hospitalized patients who met the inclusion criteria for their routine treatment. Before the procedure, the skin of the catheter insertion site was cleaned with an appropriate antiseptic solution according to the randomization groups.
  After skin cleansing, a catheter was inserted. The inserted catheters were fixed with a transparent catheter fixing tape. The introductory information section on the patient in the data collection form was filled in before the procedure, information on catheterization and catheter infection follow-up sections after the insertion of the peripheric intravenous catheter.

OTHER OUTCOMES:
Efficacy and Safety: Vital signs - Body temperature | Twelve hours, 15 minutes, 2 repeated measurements
  Effectiveness and safety in practice: After insertion of the catheters, body temperatures were observed at 12-hour intervals.
  The body temperature of the patients was measured with intratympanic degrees before the catheter was inserted and at the 12th and 24th hours after the catheter was inserted and recorded in the data collection form. Before the measurements, the child was allowed to rest for about 3-5 minutes.
Efficacy and Safety: Vital signs- Heart rate | Twelve hours, 15 minutes, 2 repeated measurements
  Effectiveness and safety in practice:
  The heart rate of the patients was measured before insertion of the catheter and at the 12th and 24th hours after the insertion of the catheter, and recorded on the data collection form, by means of the pulseeoxymeter tape using the monitor attached to the finger.
  Before the measurements, the child was allowed to rest for about 3-5 minutes.
Efficacy and Safety: Vital Signs - Blood pressure | Twelve hours, 15 minutes, 2 repeated measurements
  Effectiveness and safety in practice: After insertion of the catheters, blood pressures were observed at 12-hour intervals.
  The blood pressure of the patients was measured before the catheter was inserted and at the 12th and 24th hours after the catheter was placed, using the monitor attached to the cuff attached to the patient's arm, and recorded on the data collection form.
  measurements were made each time from the same extremity. Before the measurements, the child was allowed to rest for about 3-5 minutes.
Efficacy and Safety: Vital signs - Oxygen saturation | Twelve hours, 15 minutes, 2 repeated measurements
  Effectiveness and safety in practice: After insertion of the catheters, oxygen saturations were observed at 12-hour intervals.
  The oxygen saturations of the patients were measured before the catheter was inserted and at the 12th and 24th hours after the catheter was placed, and recorded on the data collection form, using the monitor attached to the pulseeoxymeter band attached to the fingers.
  Measurements were made on the same finger each time. Before the measurements, the child was allowed to rest for about 3-5 minutes.
Efficacy and Safety: Vital signs - Respiratory | Twelve hours, 15 minutes, 2 repeated measurements
  Effectiveness and safety in practice: After insertion of the catheters, respiratory counts were observed at 12-hour intervals.
  Respiratory rates of the patients were measured before the catheter was inserted and at the 12th and 24th hours after the catheter was inserted through the monitor connected to the electrodes attached to the patients' chest and recorded on the data collection form.
  Before the measurements, the child was allowed to rest for about 3-5 minutes.
Efficacy and Safety: Local infection - Temperature change | Twelve hours, 15 minutes, 2 repeated inspection
  Efficiency and safety in application:
  The local temperature change of the patients was measured by the investigator at the catheter insertion site at the 12th and 24th hours with a non-contact infrared thermometer. And recorded in the data collection form. All observations were made by the researcher.
Efficacy and Safety: Local infection - Discharge/drainage | Twelve hours, 15 minutes, 2 repeated inspection
  Effectiveness and safety in practice:
  The local infection findings of the patients were observed by the investigator at the 12th and 24th hours of the catheter insertion site and recorded on the data collection form.
  All observations were made by the researcher. Discharge/drainage was questioned as if there was no drainage/discharge in the patient when the catheter insertion was on sight.
  It was evaluated as either "yes" or "no".
Efficacy and Safety: Local infection - Pain | Twelve hours, 15 minutes, 2 repeated inspection
  Efficacy and safety in practice: After insertion of the catheters, the catheter insertion site was observed and asked every twelve hours for local pain.
  It was evaluated as either "yes" or "no". All observations were made by the researcher. It was recorded in the data collection form.
Efficacy and Safety: Local infection - Tenderness | Twelve hours, 15 minutes, 2 repeated inspection
  Effectiveness and safety in practice:
  The local infection findings of the patients were observed by the investigator at the 12th and 24th hours of the catheter insertion site and recorded on the data collection form.
  All observations were made by the researcher. Tenderness was questioned as if there was no sensitivity in the patient when the catheter insertion was touched.
  It was evaluated as either "yes" or "no".
Efficacy and Safety: Local infection - Swelling | Twelve hours, 15 minutes, 2 repeated inspection
  Effectiveness and safety in practice:
  The local infection findings of the patients were observed by the investigator at the 12th and 24th hours of the catheter insertion site and recorded on the data collection form.
  All observations were made by the researcher. Swelling was questioned as if there was no swelling in the patient when the catheter insertion was touched.
  It was evaluated as either "yes" or "not no".
Efficacy and Safety: Skin swab effectiveness | 5 months
  A swab sample was taken from the catheter insertion site at the 1st and 24th hours. The presence of bacterial growth at the catheter insertion site was examined. The same process was repeated 24 hours later, and the presence of growth between the two procedures was evaluated. The result of the skin swab analysis was displayed on the computer on the third day after the sample delivery, in the patient's information section. The results were recorded in the data collection form.
  After the peripheral catheter was inserted, a swab sample was taken from the cannula entrance at the 1st and 24th hours, using a sterile cotton applicator soaked in sterile distilled water, in accordance with the protocol created by scanning the literature.
  The sample taken was sent to the patient for bacterial analysis in his laboratory without waiting.
  Analysis results were recorded on the eidlip data collection form obtained from the patient results system available on the computer 3 days after each sample.
Efficacy and Safety: Laboratory analysis | 5 months
  Routine blood samples were not taken from the patients to determine the presence of systemic infection.
  Blood analysis is performed routinely in the clinic, immediately after hospitalization and at the 24th hour.
  The blood analysis at the first admission and the results of the blood analysis 24 hours later were taken from the physician files.
  According to the local infection indicators and clinical conditions of the patients, it was decided to take and send samples for blood culture upon the physician's request.
  Before the application, the results of the routine examinations sent with the request of the physician were checked.
  Complicated blood culture results, white blood cell count (WBC), C-reactive protein (CRP) level results were recorded on the data collection form.

CONTACTS AND LOCATIONS:
Overall Officials: Aysegul Simsek, PhD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Avcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After the study is published in a journal in article format, I can share it.

REFERENCES:
- [Background] Abolfotouh MA, Salam M, Bani-Mustafa A, White D, Balkhy HH. Prospective study of incidence and predictors of peripheral intravenous catheter-induced complications. Ther Clin Risk Manag. 2014 Dec 8;10:993-1001. doi: 10.2147/TCRM.S74685. eCollection 2014. PMID 25525365
- [Background] Adams D, Elliot TS. Skin antiseptics used prior to intravascular catheter insertion. Br J Nurs. 2007 Mar 8-21;16(5):278-80. doi: 10.12968/bjon.2007.16.5.22997. PMID 17505372
- [Background] Berry AM. A comparison of Listerine(R) and sodium bicarbonate oral cleansing solutions on dental plaque colonisation and incidence of ventilator associated pneumonia in mechanically ventilated patients: a randomised control trial. Intensive Crit Care Nurs. 2013 Oct;29(5):275-81. doi: 10.1016/j.iccn.2013.01.002. Epub 2013 May 19. PMID 23692975
- [Background] Bolton D. Improving peripheral cannulation practice at an NHS Trust. Br J Nurs. 2010 Nov 25-Dec 8;19(21):1346, 1348-50. doi: 10.12968/bjon.2010.19.21.79998. PMID 21355359
- [Background] Letscher-Bru V, Obszynski CM, Samsoen M, Sabou M, Waller J, Candolfi E. Antifungal activity of sodium bicarbonate against fungal agents causing superficial infections. Mycopathologia. 2013 Feb;175(1-2):153-8. doi: 10.1007/s11046-012-9583-2. Epub 2012 Sep 19. PMID 22991095
- [Background] Ding L, Wu HL, Zhu JH, Ding M, Wang YL, Xu XJ. Superiority of 5% NaHCO3 for preoperative hair removal in patients undergoing coronary artery bypass graft surgery with a limb vein: a randomized controlled trialdagger. Eur J Cardiothorac Surg. 2014 Aug;46(2):e28-32. doi: 10.1093/ejcts/ezu203. Epub 2014 Jun 18. PMID 24948414
- [Background] Wu HL, Xu YH, Shi JH. 5% NaHCO3 Is Appropriate for Skin Cleaning With Central Venous Catheters. Am J Med Sci. 2017 Jan;353(1):12-16. doi: 10.1016/j.amjms.2016.10.010. Epub 2016 Oct 29. PMID 28104097
- See also: Adıgüzel, Ö. (2015). Klorheksidin. Turkiye Klinikleri J Endod-Special Topics, 1(2), 15-9. — https://www.turkiyeklinikleri.com/article/tr-klorheksidin-72909.html
- See also: Aktaş, E., Sarı, E.N., Seremet Keskin, A., Pişkin, N., Külah, C., Cömert, F. (2011) Damar İçi Kateter ile İlişkili Enfeksiyon Etkenleri ve Antibiyotik Duyarlılıkları. Mikrobiyoloji Bülteni, 45(1), 86-92. — http://www.mikrobiyolbul.org/managete/fu_folder/2011-01/html/2011-45-01-086-092.htm
- See also: 12. Centers for Disease Control and Prevention (CDC), (2002). CDC Guideline for the Prevention of Intravascular Catheter-Related Infections. MMWR August 9, 2002. (37) — https://www.cdc.gov/mmwr/preview/mmwrhtml/rr5110a1.htm